CLINICAL TRIAL: NCT02460367
Title: A Phase 1b/2 Study of Tergenpumatucel-L (HyperAcute Lung) Immunotherapy in Combination With the IDO Pathway Inhibitor Indoximod and Docetaxel in Patients With Advanced Previously Treated Non-Small Cell Lung Cancer (NSCLS)
Brief Title: Immunotherapy Combination Study in Advanced Previously Treated Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment and changing landscape of standard of care.
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0401; 1504-1393 (Other: Office of Biotechnology Activities)
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer; Progression of Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Recurrent
Keywords: Non-small Cell Lung Cancer; Vaccine Therapy; Immunotherapy; Second line therapy; Progressive; Relapsed; IDO; IDO Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Docetaxel; 1-methyltryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1: Dose Escalation (Experimental): Up to 18 participants will be enrolled and treated at escalating doses of Indoximod with a fixed dose of tergenpumatucel-L and docetaxel. Treatment may continue until definitive disease progression or significant toxicology.
  Interventions: Drug: Docetaxel; Biological: Tergenpumatucel-L; Drug: Indoximod

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere®
Biological: Tergenpumatucel-L
  Other Names: HyperAcute®-Lung Immunotherapy
Drug: Indoximod
  Other Names: D-1MT; 1-methyl-D-tryptophan

SUMMARY:
This is a Phase 1/2 trial using indoximod, an inhibitor of the immune "checkpoint" pathway indoleamine 2,3-dioxygenase (IDO), in combination with Tergenpumatucel-L immunotherapy and Docetaxel to treat subjects with advanced Non-Small Cell Lung Cancer (NSCLC). From a practical standpoint, a successful tumor immunotherapy will likely require a combination treatment with additional therapeutic interventions that both activate an immune response and remove redundant mechanisms of tolerance maintenance. This clinical trial utilizes the combination of the chemotherapeutic agent, docetaxel, plus two investigational methods of cancer immunotherapy: the first, tergenpumatucel-L, is intended to educate the human immune system to recognize the abnormal components found in lung cancer cells, resulting in an immune response intended to destroy or block the growth of the cancer; and the second, the IDO inhibitor Indoximod, will overcome tumor-induced immune suppression.

The goal of this study is to assess the progression-free survival (PFS) and overall survival (OS) rates in this patient population. This study will provide a foundation for future trials testing indoximod combined with tergenpumatucel-L.

ELIGIBILITY:
Inclusion Criteria

* Histological/cytological diagnosis of non-small cell lung cancer (NSCLC). Squamous cell (epidermoid), adenocarcinoma, bronchoalveolar carcinoma and large cell anaplastic lung carcinoma histologies are eligible. Mixed histologies of NSCLC (i.e., adenosquamous) are eligible. Mixed NSCLC/small cell lung carcinoma (SCLC), and variant large and small cell lung cancer are NOT eligible for this study.
* Measurable disease as defined by RECIST 1.1 Criteria.
* At least one but no more than three prior lines of therapy in the advanced stage are allowed. One prior line of therapy must be platinum doublet chemotherapy.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Marrow: Hemoglobin ≥10.0 gm/dL, absolute granulocyte count (AGC) ≥1,000/mm3 platelets ≥100,000/mm3, absolute lymphocyte count ≥1000/mm3.
  * Hepatic: Serum/plasma total bilirubin ≤1.5 x upper limit of normal (ULN) with the exception of <2.9 mg/dL for patients with Gilbert's disease, ALT (SGPT) and AST (SGOT) ≤2.5 x ULN.
  * Renal: Serum/plasma creatinine (sCr) ≤1.5 x upper limit of normal, or creatinine clearance (Ccr) ≥50 mL/min.
* Serum/plasma albumin > 3.0 gm/dL
* Sexually active women of child-bearing potential must agree to use two forms of contraception prior to study entry and for the duration of study participation. A pregnancy test is required prior to study enrollment and monthly while on treatment with indoximod for all women of child- bearing potential. Also men should be discouraged from fathering children while on treatment.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria

* More than three lines of prior therapy.
* Previous use of indoximod or tergenpumatucel-L immunotherapy.
* A history of other malignancy, unless treated with curative intent, and no evidence of disease for at least 2 years.
* Current therapy with any other investigational agents.
* Untreated CNS disease, metastases or carcinomatous meningitis. Patients with CNS metastases must be at least 2 weeks status post prior therapy to the brain and be off all steroids without progressing CNS disease or symptoms.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to indoximod, docetaxel, or other agents used in the study.
* Current use of immunosuppressive drugs or use of corticosteroids, except for inhaler, topical corticosteroids, or dexamethasone in the premedication for docetaxel.
* Other malignancy within three years, unless the probability of recurrence of the prior malignancy is <5%. Patient's curatively treated for squamous cell carcinoma and basal cell carcinoma of the skin and carcinoma in situ of the uterine cervix (CIN) or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant.
* Any of the following within 6 months prior to study drug administration:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled ongoing cardiac dysrhythmias of ≥ grade 2, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the unknown potential for pharmacokinetic interactions with indoximod, or docetaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy.
* Active autoimmune disease requiring systemic therapy. Patients with a history of autoimmune disease must be counselled regarding the unknown potential of exacerbating or reactivating previous or dormant autoimmunity during the consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07-17 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Regimen Limiting Toxicity | Approximately 6 weeks
  Phase 1 component: To identify the regimen limiting toxicity (RLT) for the combination of tergenpumatucel-L and indoximod.
Progression Free Survival (PFS) | Approximately 18 months

SECONDARY OUTCOMES:
Frequency and grade of adverse events of tergenpumatuucel-L, indoximod and docetaxel | Approximately 18 months
Objective Response Rate | Approximately 18 months
  To assess preliminary evidence of efficacy of tergenpumatuucel-L, indoximod and docetaxel using RECIST 1.1 measurement criteria.
Overall Survival | Approximately 30 months
Response rate to subsequent therapy | up to 36 months
  Assess evidence of delayed response of tergenpumatuucel-L, indoximod and docetaxel using RECIST 1.1 measurement criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gene Kennedy, MD, Study Director — NewLink Genetics Corporation
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No